CLINICAL TRIAL: NCT06965192
Title: Designing Visual Tools to Enhance Cancer Surgeon Decision-making
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: LCC2321Aim3
Record Dates: First submitted 2025-05-01; First posted 2025-05-11 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer; Kidney Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient participants (Experimental): Patient participants will complete a 10-minute baseline survey, 15-minute after-visit survey and 5-minute 6-month survey.
  Interventions: Other: No intervention
- Physician participants (Experimental): Physician participants seeing patients with newly diagnosed localized prostate cancer and clinical T1 renal masses suspicious for kidney cancer.
  Interventions: Behavioral: Visual

INTERVENTIONS:
Behavioral: Visual — Physician participants will view the visual decision support before entering the patient's room during the intervention period, with the option to share with the patient.
  Arms: Physician participants
Other: No intervention — No intervention
  Arms: Patient participants

SUMMARY:
This prospective study will compare pre-post pilot test of surgeon-facing, visual decision support among urologists seeing patients with newly diagnosed localized prostate and kidney cancer. Up to 20 urologists (10 academic and 10 community) will be enrolled. The goal will be to capture up to 10 pre- and 10 post-intervention patient encounters for each urologist with an accrual target of 200 unique patient visits (100 pre and 100 post-intervention) over a half-year period. Patient encounters pre- and post-intervention will be audio recorded, transcribed, and coded for discussion of risks/benefits of surgery and strength of recommendation. Patients and urologists will complete additional surveys on their perceptions of patient-provider communication. Urologists will further describe their experience and rate their satisfaction with visual decision support. Communication (content and perceived) will be compared pre- and post-intervention with secondary comparisons by race and care setting.

It was hypothesized that the discussion of risks and benefits of cancer surgery will increase post-intervention and that the strength of recommendation and perceptions of patient-provider communication will change. The secondary hypothesis is that these changes will differ by patient race and care setting.

ELIGIBILITY:
Inclusion Criteria:

In order to participate in this study, a subject must meet all of the eligibility criteria outlined below.

* Verbal informed consent was obtained to participate in the study.
* Subject is willing and able to comply with study procedures based on the judgment of the investigator or protocol designee.
* Age ≥ 18 years at the time of consent.
* For patient subjects, HIPAA authorization for the release of personal health information and a new histologic diagnosis of localized prostate cancer based on prostate biopsy or clinical diagnosis of T1 renal mass (≤7 cm in diameter) Suspicion for kidney cancer based on cross-sectional imaging. New diagnosis is defined as within 6 months of consent. T1 renal masses include solid masses or Bosniak III/IV cystic masses.
* For physician subjects, practicing urologist in North Carolina at UNC Health, Novant Health, or an affiliated site and sees patients with suspected or confirmed prostate or kidney cancer.

Exclusion Criteria:

The subjects meeting the following criteria will be excluded from study participation:

* Non-English speaking.
* Unwilling or unable to complete informed consent.
* For patient subjects:

  1. Has staging information indicating locally advanced or metastatic disease. This would include PSA >50 ng/ml, imaging suggestive of distant metastasis, or lymph node involvement, renal masses >7 cm or invading in renal sinus or tumor thrombus.
  2. Histologic or clinical diagnosis >6 months before date of consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Discussion of Risks and Benefits | Baseline (Patient-Physician Encounter)
  The impact of visual decision support on patient-physician communication will be assessed using coding-based thematic analysis of the debriefing interviews. The Informed Decision-Making coding system, which includes 9 elements which includes the nature of the clinical problem (e.g., cancer mortality risk, life expectancy), treatment options (e.g., surgery, alternatives), risks and benefits (e.g., complications, side effects, functional outcomes), and uncertainties (e.g., range of possible outcomes). Audio-recorded patient encounters will be coded. Paired coders will score these domains as a 0 (absent), 1 (partial, brief, or one-way), or 2 (complete, two-way discussion).

SECONDARY OUTCOMES:
The impact of the visual decision support on the strength of the recommendations - observer | Baseline (Patient-Physician Encounter)
  The impact of the visual decision support on the strength of the recommendations will be assessed using coding-based thematic analysis of the debriefing interviews. An established coding approach is applied to audio-recorded patient encounters. Recommendations for surgery will be rated by paired coders from -2 to +2, with ±2 being strong, ±1 being mild, and 0 being neutral. To compare the impact of the visual decision support on communication, patient decision-making, physician decision-making, and treatment selection/quality.
The impact of the visual decision support on the strength of the recommendations - surgeon rated | Baseline (After-Visit)
  Surgeon participants will rate the strength of recommendation after each patient visit on a 5-point Likert scale with 1 being strong against surgery, 5 being strong for surgery, and 3 being neutral.
Patient-Centered Communication | Baseline (After-Visit)
  Patient-Centered Communication in Cancer will be assessed using 6-item validated scale on patient perspective of communication that incorporates questions on exchanging information, fostering relationships, making decisions, responding to emotions, enabling self-efficacy, and managing uncertainty. Maximum value=5, Minimum value=1; higher score means better outcome.
Physician Satisfaction Scale | Baseline (After-Visit)
  Physician Satisfaction Scale will be assessed using the 3-item scale on physician perception of the quality of the consultation and patient's understanding of their case and treatment options. Maximum value=5, Minimum value=1; higher score means better outcome.
Patient-Physician Communication | Baseline (After-Visit)
  Patient-Physician Communication will be assessed using the 1 subscale (5 items) on each surgeon's "contextual knowledge of the patient" as perceived by the patient. Maximum value=5, Minimum value=1; higher score means better outcome.
Patient Decision-Making | Up to 6 months
  Patient Decision-Making includes shared decision-making, knowledge, and trust in surgical decision, decisional conflict, decisional regret, and self-efficacy will be assessed using questionnaire.
  * Decisional conflict - max 100, min 0, lower score is better
  * Decisional regret - max 100, min 0, lower score is better
  * Trust - max 5, min 1, higher score better
  * Shared Decision Making Questionnaire (SDM-Q-9) - max 45, min 0, higher score is better
  * Self-Efficacy - max 5, min 1, higher score better
Physician Decision-Making | Baseline (After-Visit)
  Physician Decision-Making includes perceived risk, recommendations for surgery, and whether they shared the visual decision support with the patient during the visit will be assessed.
  * Risk perception (0-100)
  * Surgery Rating (1-5)
Treatment Selection/Quality | Up to12 months
  Treatment Selection/Quality includes Choice of surgery (including type), Observation (including active surveillance, watchful waiting), Other treatment (e.g., radiationtherapy, ablative treatment), ancillary testing (e.g., receipt of biomarker,see condary imaging, renal mass biopsy, outside referral).
Perceived Usability Ratings | Up to 6 months
  Perceived Usability Ratings, including Ratings on acceptability, appropriateness, feasibility, usefulness, supportiveness, informativeness, aesthetics, and ease of use will be assessed.
  Maximum value=5, Minimum value=1; higher score means better outcome.
Physician Debriefing Interview | Up to 6 months
  Physician Debriefing Interview will be assessed with a study-specific interview guide. Participants will be asked for their subjective assessment of perceived usefulness, ease of use, workflow impact, and overall satisfaction. Barriers to use and suggestions for improvements will also be elicited

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Jui Tan, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (2):
- United States (2):
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - New Hanover Regional Medical Center, Wilmington, North Carolina

IPD SHARING:
Plan to Share IPD: No
The data will be made available upon reasonable request.

REFERENCES:
- See also: Clinical trials at UNC Lineberger — http://unclineberger.org/patientcare/clinical-trials/clinical-trials